CLINICAL TRIAL: NCT01461512
Title: The Effects of Intravenous Heme Arginate on Functional Magnetic Resonance Imaging During Ischemia
Brief Title: Heme Arginate in Functional Magnetic Resonance Imaging (fMRI)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: MWolzt (Other)
Responsible Party: Sponsor-Investigator, MWolzt, Prof. Dr. Michael Wolzt, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Version 1.2 2008-006967-35
Record Dates: First submitted 2011-10-14; First posted 2011-10-28 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2011-10

CONDITIONS: Ischemia-reperfusion Injury
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo administration
- Heme arginate treatment (Experimental)
  Interventions: Drug: heme arginate administration

INTERVENTIONS:
Drug: heme arginate administration — heme arginate 1 mg/kg body weight 24 hours prior to ischemia
  Arms: Heme arginate treatment
Drug: Placebo administration — NaCl isotonic
  Arms: Placebo

SUMMARY:
Ischemia reperfusion injury may be attenuated by HO-1 induction. Heme arginate showed protective effects during prolonged ischemia in animal studies. Functional blood oxygen level dependent (BOLD) magnetic resonance imaging (MRI) shall evaluate the effects of HO-1 induction during short-time ischemia in skeletal muscle of healthy subjects.

DETAILED DESCRIPTION:
Ischemia reperfusion injury may be attenuated by HO-1 induction. Heme arginate showed protective effects during prolonged ischemia in animal studies. The investigators previous data confirmed strong HO-1 induction following heme arginate infusion in healthy humans. Therefore, the investigators next approach is to evaluate the direct effects of heme arginate on short time Ischemia-reperfusion (IR) injury in healthy humans. This will be done by the following surrogate markers of IR injury.

Functional blood oxygen level dependent (BOLD) magnetic resonance imaging (MRI) can measure alterations in tissue oxygenation in a high spatial and temporal resolution. This non-invasive methods therefore represent a promising technique to evaluate the effects of HO-1 induction on energy metabolism and oxygen saturation during ischemic stress and short time reperfusion in skeletal muscle.

As additional outcome, levels of myoglobin and creatine-kinase will be measured in plasma according to standard laboratory procedures.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Men aged between 18 and 46 years (inclusive)
* Nonsmoker for more than 3 months
* Body mass index between 18 and 27 kg/m2
* Normal findings in medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Negative results from urine drug screen if performed
* Ability to communicate well with the investigator in the local language and to understand and comply with the requirements of the study

Exclusion Criteria:

* Known hypersensitivity to the study drug or any excipients of the drug formulation
* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment with another investigational drug within 3 weeks prior to screening
* History or clinical evidence of any disease and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism or excretion of the study drug
* Evidence of hypertension, pathologic hyperglycemia, hyperlipidemia
* Treatment in the previous 3 weeks with any drug including over-the-counter drugs (including herbal medicines such as St John's Wort)
* Symptoms of a clinically relevant illness in the 2 weeks before the first study day
* Blood donation during the previous 3 weeks
* Any metallic, electric, electronic or magnetic device or object not removable
* Claustrophobia

Ages: 18 Years to 46 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-01; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
BOLD MRI signal | 2 minutes prior to ischemia till 25 minutes after ischemia
  functional MRI assessment of blood oxygen level dependent signal strength
Serum markers of myocellular injury | 24 hours after ischemia
  (myoglobin, creatine-kinase)

SECONDARY OUTCOMES:
Blood pressure | 20 minutes prior to and 40 minutes after ischemia
  in mmHg
Heart rate | prior to and after ischemia
  in beats per minute

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Department of Clinical Pharmacology, Vienna, Austria

REFERENCES:
- [Derived] Andreas M, Schmid AI, Doberer D, Schewzow K, Weisshaar S, Heinze G, Bilban M, Moser E, Wolzt M. Heme arginate improves reperfusion patterns after ischemia: a randomized, placebo-controlled trial in healthy male subjects. J Cardiovasc Magn Reson. 2012 Aug 2;14(1):55. doi: 10.1186/1532-429X-14-55. PMID 22857721